CLINICAL TRIAL: NCT03587220
Title: En undersøgelse af Mekanismerne Bag Nociceptiv Desensibilisering forårsaget af Topikal Capsaicin
Brief Title: A Mechanistic Evaluation of the Nociceptive Desensitizing Properties of Topical Capsaicin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Biologist, PhD, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20180034
Record Dates: First submitted 2018-06-21; First posted 2018-07-16 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Capsaicin; Ultaviolet B Light Burn; Neuropathic Pain; Lidocaine
MeSH Terms: conditions — Neuralgia | interventions — Capsaicin; Radiation; Tumor Protein, Translationally-Controlled 1; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsaicin+UVB group (Experimental): All subjects will be treated with capsaicin, placebo + UVB, or Capsaicin+UVB.
  Interventions: Drug: Capsaicin Topical; Radiation: Ultraviolet-B (UVB) irradiation
- Capsaicin + EMLA group (Experimental): All subjects will be pre-treated with lidocain cream before capsaicin application
  Interventions: Drug: Capsaicin Topical; Other: Histamine 1%; Drug: Lidocaine

INTERVENTIONS:
Drug: Capsaicin Topical — Capsaicin patches (dosage form: patch 8% Qutenza) will be applied on 4x4 cm squared areas on the volar forearm. The patches will be left in place for 24h and 3 hours after which they will be removed.
Radiation: Ultraviolet-B (UVB) irradiation — Two circular areas (Ø 2 cm) on the forearm are irradiated with 2 x MED (Minimal Erythema Dose) dose of UVB using a calibrated UVB machine (290-320nm wavelength), Saal Mann Multi Tester (Mann Saal, LT SBC 400 Herford, Germany).
  Arms: Capsaicin+UVB group
Other: Histamine 1% — To deliver histamine, standard allergy skin prick test (SPT) lancets are applied. The lancets have a 1 mm shouldered tip adapt to introduce a small amount of test substance extremely locally and approximately at the dermo-epidermal junction.
  Arms: Capsaicin + EMLA group
Drug: Lidocaine — Cutaneous anaesthesia will be topically induced by using EMLA cream 5%, a local anaesthetic cream consisting of equal parts of lidocaine and prilocaine (1g contains 25 mg of lidocaine and 25 mg of prilocaine)
  Arms: Capsaicin + EMLA group

SUMMARY:
The aim of this project is to study the role of transient receptor potential (TRP-) channel V1 (TRPV1+) fibers in the development of cutaneous inflammation induced by epidermal Ultraviolet-B damage. Moreover, in this project the investigators want to evaluate if the capsaicin-desensitization action can still be induced in a skin area pretreated with topical, local anesthetic lidocaine.

DETAILED DESCRIPTION:
In this project the Ultraviolet- B pain model, a model using type B ultraviolet rays to induce a first-degree sunburn, will be used to induce a non-specific inflammation in the skin. This model is well-known to produce both peripheral and central hyperalgesia through sensitization of peripheral and central nociceptors. Capsaicin, the active substance in chili peppers, is currently used to treat peripheral neuropathic pain, and prolonged application of 8% capsaicin patch causes profound desensitization to painful heat stimuli and itch provocations. Therefore, the investigators would like to monitor the development of unspecific UVB-cutaneous inflammation and consequent neurogenic flare in a capsaicin pre-treated area. Moreover the investigators want to test if pre-treating the skin with lidocaine can reduce the pain associated with the capsaicin application without affecting its desensitization action.

ELIGIBILITY:
Inclusion criteria:

* Healthy men and women
* 18-60 years
* Caucasian descent (only in sub-study 1)
* Speak and understand English

Exclusion criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids or other drugs
* Previous or current neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate
* Current use of medications that may affect the trial
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Moles or tattoos in the area to be treated or tested.
* Exposure of the irradiated area to UV radiation (e.g., sun) 48 hours before the study days and between these
* Acute or chronic pain
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical trials)
* Known history of anaphylactic shock, or local allergy (contact dermatitis) to lidocaine, prilocaine or other local anaesthetics of the amide type.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Superficial blood perfusion measured by a Speckle contrast imager (FLPI, Moor Instruments, England). | Changes from baseline to 7 days after intervention
Measurement of Warm Detection Thresholds and Heat thresholds by using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. | Changes from baseline to 7 days after intervention
Measurement of Pain to Supra-threshold Heat Stimuli by using a PATHWAY ATS (Medoc Ltd, Israel) thermal sensory testing device. | Changes from baseline to 7 days after intervention
Measurement of Mechanical Pain Thresholds and Sensitivity using a pin-prick set consisting of 8 needles each having a diameter of 0.6 mm and different force applications: 0.8, 1.6, 3.2, 6.4, 12.8, 25.6, 50.1 and 60.0 g. | Changes from baseline to 7 days after intervention
Trans-epidermal Water Loss (TEWL) using a 2x2 cm probe to measure the humidity gradient of the skin. | Changes from baseline to 7 days after intervention

SECONDARY OUTCOMES:
assessment of pain rating by using a visual analog scales (VAS) | Change from baseline to 24 h
  The subject will report the peak and average of the perceived pain sensation during the last 24 hours (on a VAs scale from 0 indicating 'no pain' to100 indicating 'worst imaginable pain').
Itch rating by using a visual analog scales (VAS) | Changes from baseline to 7 days after intervention
  Itch is monitored for 9 minutes using a visual analog scale from 0 indicating 'no itch' to100 indicating 'worst imaginable itch.

CONTACTS AND LOCATIONS:
Locations (1):
- Silvia Lo Vecchio, Aalborg, North Denmark, Denmark